CLINICAL TRIAL: NCT01992289
Title: Extension Study of XLHED-Affected Male Subjects Treated With EDI200 in Protocol ECP-002
Acronym: ECP-002e
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Edimer Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: ECP-002e; 1R01FD005099-01 (FDA)
Record Dates: First submitted 2013-11-12; First posted 2013-11-25 (Estimated); Last update posted 2017-09-05 (Actual); Status verified 2017-08

CONDITIONS: X-linked Hypohidrotic Ectodermal Dysplasia
Keywords: XLHED; HED; Hypohidrotic ectodermal dysplasia; Christ-Siemens-Touraine Syndrome
MeSH Terms: conditions — Ectodermal Dysplasia 1, Anhidrotic | interventions — Fc-EDA

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- No treatment: This is a long-term follow-up study of subjects that received EDI200 as part of protocol ECP-002.
  Interventions: Drug: EDI200

INTERVENTIONS:
Drug: EDI200 — Long-term follow-up study of subjects that received EDI200 as part of protocol ECP-002
  Other Names: APO200

SUMMARY:
The goal of the ECP-002e extension study is to continue the evaluation of all EDI200-treated ECP-002 subjects up to age 10 yrs. No additional study drug administration is planned. The efficacy evaluations will incorporate growth and development parameters, frequency of infections and hospitalizations, and age-appropriate assessments of ectoderm-derived organ function. The safety evaluations will include physical examinations, adverse events and concomitant medication documentation, and laboratory testing. Funding Source - FDA OOPD

DETAILED DESCRIPTION:
X-linked hypohidrotic ectodermal dysplasia (XLHED) is a disorder of ectoderm development in which sweat and other secretory gland hypoplasias predispose affected infants to serious and potentially life-threatening hyperthermia and pneumonia. Those XLHED patients who survive infancy face a host of ectoderm-related clinical conditions including failure to thrive, oligodontia and misshapen teeth, mid-face hypoplasia, eczema, chronic dry eyes, asthma, respiratory infections, sinusitis and chronic nosebleeds. XLHED is caused by inherited defects in the ectodysplasin gene (EDA, www.ncbi.nlm.nih.gov/omim) resulting in a deficiency of the ectoderm signaling protein EDA-A1. As is the general case with X-linked disorders, hemizygous XLHED males are more consistently and severely affected, while heterozygous XLHED females have a more variable phenotype.

In normal development, EDA-A1 acts as an ectoderm signaling molecule that binds specifically to the EDA-A1 receptor (EDAR) triggering initiation and maturation of ectodermal appendages into sweat and other secretory glands, tooth buds and hair follicles. In the case of XLHED, EDA-A1 deficiency results in the absence or functional hypoplasia of the ectoderm appendages. There are no therapies currently available for XLHED that prevent or correct the underlying ectodermal abnormalities.

EDI200 is a fully humanized EDA-A1 replacement molecule under development as a novel therapeutic for XLHED. EDI200 comprises the human IgG1 Fc domain linked to the human EDA-A1 receptor-binding domain. On-target EDI200 activation of the EDA-A1/EDAR signaling pathway in vivo is evidenced by the remarkable phenotypic response in preclinical models. In XLHED-affected animals, EDA-A1 deficiency is corrected by a single course of EDI200 therapy, administered either prenatally (mice) or postnatally (newborn mice and dogs), resulting in a significant and sustained improvement in the health of the treated animals. Postnatal studies in both mice and dogs demonstrated a consistent and restricted window of efficacy. These results support the clinical development of EDI200 as a therapeutic to be administered to XLHED-affected patients in the neonatal period or earlier.

ECP-002, a Phase 2, international, first-in-neonate EDI200 study is enrolling treatment-naïve, XLHED-affected male newborns in the first two weeks of life. All subjects will meet entry criteria including documentation of an EDA mutation associated with XLHED. Following Baseline evaluations, EDI200 dosing is initiated between day-of-life 2 and 14, with each study subject receiving a single course of study drug administered at 2 doses/week for a total of 5 doses. The treatment study protocol incorporates comprehensive safety, pharmacokinetic (PK), immunogenetic, and pharmacodynamic (PD)/efficacy evaluations continuing through age 6 months.

The goal of the ECP-002e extension study is to continue the evaluation of all EDI200-treated ECP-002 subjects up to age 10 yrs. No additional study drug administration is planned. The efficacy evaluations will incorporate growth and development parameters, frequency of infections and hospitalizations, and age-appropriate assessments of ectoderm-derived organ function. The safety evaluations will include physical examinations, adverse events and concomitant medication documentation, and laboratory testing.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following criteria to be enrolled:

1. Subject received at least one dose of EDI200 in the neonate study ECP-002
2. Written informed consent of parent(s)

Exclusion Criteria:

Subjects who meet any of the following criteria may not be enrolled in this study:

1. Medically-significant postnatal complications or congenital anomalies outside of those considered to be associated with the diagnosis of XLHED
2. Major protocol violations during enrollment in study ECP-002 as determined by the Sponsor

Ages: 6 Months to 1 Year | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Study Population: This is an open-label extension study without additional study drug administration on as many as 10 XLHED-affected males previously having received EDI200 in the ECP-002 trial. XLHED-affected male infants who completed the ECP-002 trial will be followed with yearly visits starting at age 1 year.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2014-03; Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Growth and development | Annually up to age 10 years
  Growth and development as compared with age-matched standards
Dentition | Change from baseline dentition at 2, 5 and 10 years
  Dentition assessed by dental examinations and radiographs at ages 2 yrs, 5 yrs, and 10 yrs

SECONDARY OUTCOMES:
Mortality | Annually up to age 10 years
  At each annual visit the subject and his family will be questioned regarding mortality, hospitalization, infections, unexplained fevers and heat intolerance occurring since the last annual visit.
Hospitalizations | Annually up to age 10 years
  At each annual visit the subject and his family will be questioned regarding mortality, hospitalization, infections, unexplained fevers and heat intolerance occurring since the last annual visit.
Infections | Annually up to age 10 years
  At each annual visit the subject and his family will be questioned regarding mortality, hospitalization, infections, unexplained fevers and heat intolerance occurring since the last annual visit.
Unexplained fevers | Annually up to age 10 years
  At each annual visit the subject and his family will be questioned regarding mortality, hospitalization, infections, unexplained fevers and heat intolerance occurring since the last annual visit.
Heat intolerance | Annually up to age 10 years
  At each annual visit the subject and his family will be questioned regarding mortality, hospitalization, infections, unexplained fevers and heat intolerance occurring since the last annual visit.
Sweat gland density | Annually up to age 10 years
  Sweat duct density (number/cm2) from at least two different sites on the soles of the feet or the palms of the hands will be determined through analysis of images collected annually if positive findings were observed at the end of protocol ECP-002 and will continue until negative results are observed on two consecutive evaluations. This will be accomplished by direct visualization with an FDA 510(k) device, the Lucid VivaScope 1500 (www.lucid-tech.com). This technology has been tested in controls and XLHED-affected males from the newborn period to adulthood without complication. An adhesive ring will be placed on the subject's palm to which the VivaScope will be attached via a magnetic lock. A series of photographs will be taken of an area approximately 6mm X 6mm. An individual trained in the use of this device will be involved in the acquisition of all images.
Sweat function | Annually up to age 10 years
  Maximal sweating on the volar lower arm surface of each subject will be induced by pilocarpine iontophoresis followed by sweat collection using the Macroduct Sweat Collection System developed primarily for sweat collection and analysis in the diagnosis of Cystic Fibrosis from the newborn period on (www.wescor.com).
  Following completion of the pilocarpine iontophoresis the Webster Sweat Inducer electrodes and discs are removed from the subject, the application site is wiped once with alcohol, and a Macroduct Sweat Collector is placed over the site of one electrode. The Macroduct Sweat Collector is held in place for approximately 30 minutes using a Velcro Macroduct Strap. Sweat volume is determined from microliter markings on a collection coil diagram. Sweat rate will be determined annually if positive findings were observed at the end of protocol ECP-002 and will continue until negative results are observed on two consecutive evaluations.
Skin health | Annually up to age 10 years
  Skin examination and history of skin disorders will be evaluated at each annual visit by detailed physical exam and medical history.
Hair growth | Change from baseline hair growth at 5 and 10 years
  At the year 5 and 10 visits the total and anagen hair counts and follicular unit counts in the scalp will be determined from color macrophotographs of clipped hair in a 1 cm2 circular target area centered by a cosmetic ink dot. Hair in the target area will first be clipped to approximately a 1 mm length for determination of total hair count and hairs per follicular unit, and then clipped further to about 0.35 mm to monitor hair growth over the 2-3 day period between phototrichograms. The sponsor will provide all of the equipment necessary for photography and to cut the hair to the exact lengths specified. A second photogram will be taken approximately 2-3 days later for the determination of anagen and telogen hair counts, based on the number of hairs that have lengthened over the intervening time period, as well as hair properties including growth rate and hair width.
Respiratory health | Annually up to age 10 years
  Annual medical history and physical exam related to asthma, sinusitis, nosebleeds and nasal congestion will be evaluated annually. Pulmonary function testing (FVC and FEV1) will be performed on all subjects starting at age 5 years at a laboratory experienced with pediatric subjects. Additionally, levels of exhaled nitric oxide (eNO) as an indicator of pulmonary inflammation will be quantified non-invasively with an age-group appropriate device in all subjects age 5 years and older.
Ocular health | Annually up to age 10 years
  The eye examination will be performed by an ophthalmologist experienced in assessments of tear film and ocular surface in infants as well as children and adults. The examination will document the presence/absence of signs of infection, inflammation and corneal irritation, as well as a tear film break-up time. For children 5 years or older the assessment will also include the Shirmer test for rate of tear production and the OCULAR SURFACE DISEASE INDEX© questionnaire.
Number of participants with adverse events | Annually up to age 10 years
  The annual safety evaluations will consist of safety laboratory sampling, assessment of adverse events and concomitant medications, and a physical examination with vital signs.

OTHER OUTCOMES:
Craniofacial development | Annually up to age 10 years
  A craniofacial recognition software algorithm is under development that will identify characteristics of XLHED-affected males as neonates, children and adults. The algorithm uses non-invasive 2D frontal photographs and will be used in this study to document changes in craniofacial appearance over time. Digital images will be obtained annually with a commercial camera, and all photographs will be anonymized (subject ID only) prior to transmission for analysis to FDNA, the company developing the software algorithm (http://www.fdna.com).
Exercise thermoregulation | Change from baseline exercise thermoregulation at 7, 8, 9 or 10 years (done once)
  Exercise thermoregulation during bicycle ergometry will be assessed once at a single visit when the study subject has reached an age of at least 7 yrs and a weight of at least 80 lbs. The main outcome measure is body core temperature during and after exercise. Body core temperature is measured immediately prior to and 4, 8, 12, 16, 20, 24, 30, 40, 60 and 90 minutes after initiation of exercise using an ingestible thermometer pill. External recording of body core temperature is started approximately 30 minutes after ingestion of a calibrated pill. Basal values are noted when no changes of body temperature is observed anymore, and the subject is then told to start cycling. Heart rate is monitored continuously. Physical strain is 0.5 W/kg body weight at the beginning and increased every 4 minutes by 0.5 W/kg body weight. Stopping criteria are a body core temperature of more than 40°C, an increase in heart rate above an age-adjusted threshold, or subjective exhaustion.
Immunogenicity | Change from baseline immunogenicity at 2 years
  Immunogenicity testing at 2 yrs of age will be compared with the results from the ECP-002 study

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Huttner, MD, PhD, Study Director — Edimer Pharmaceuticals
Locations (7):
- United States (3):
  - University of California, San Francisco, San Francisco, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Washington University School of Medicine, St Louis, Missouri
- Hôpital Necker-Enfants Malades, Paris, France
- Universitätsklinikum Erlangen, Erlangen, Bavaria, Germany
- Azienda Ospedaliera-Polo Universitario "Luigi Sacco", Milan, Italy
- University Hospital of Wales, Cardiff, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided